CLINICAL TRIAL: NCT00002353
Title: A Phase I Safety and Immunogenicity Trial of UBI HIV Lipopeptide Immunotherapeutic P3C541b in HIV-1 Seropositive Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: United Biomedical (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 090; V103B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-07

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; AIDS Vaccines
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Biological: P3C541b Lipopeptide

SUMMARY:
To evaluate an HIV lipopeptide immunotherapeutic, P3C541b, at two dose levels administered subcutaneously in HIV-seropositive patients.

DETAILED DESCRIPTION:
Patients are randomized to receive P3C541b or placebo within each of two study groups. Enrollment in the first group will be independent of HLA type, whereas all but two of the patients enrolled in group 2 must have one or more HLA types A33, B8, B27, or Bw62. Treatment in group 2 will not begin until those in group 1 have reached day 14 without serious toxicity.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV positivity.
* CD4 count >= 500 cells/mm3.
* No evidence of AIDS, persistent diarrhea, fever, oral hairy leukoplakia, herpes varicella-zoster (multidermatomal), oral candidiasis, opportunistic infections, severe cytomegalovirus infection, or disseminated or chronic herpes simplex.
* Successful establishment of EBV transformed B lymphoblastoid cell line.

NOTE:

* Most patients in group 2 must possess one or more HLA types A33, B8, B27, or Bw62.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Active syphilis.
* Positive circulating hepatitis B virus antigen.
* Active clinically significant medical problems.
* Evidence of psychiatric, medical, or substance abuse problems that would affect ability to participate on study.
* Occupational or other responsibilities that would prevent completion of study.

Concurrent Medication:

Excluded:

* Other HIV immunotherapeutic.
* Zidovudine or analog.
* Investigational therapies for HIV.

Patients with the following prior conditions are excluded:

* History of cancer unless surgically excised with reasonable assurance of cure.
* History of anaphylaxis or other serious adverse reactions to vaccines.
* History of serious allergic reaction to any substance that required hospitalization or emergent medical care (e.g., Stevens-Johnson syndrome, bronchospasms, or hypotension).
* History of autoimmune disease or use of immunosuppressive medications.
* History of suicide attempts or past psychosis.

Prior Medication:

Excluded within the past 6 months:

* HIV immunotherapeutic.
* Zidovudine or analog.
* Investigational therapies for HIV. Illicit drug use within past 30 days.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Hosp, Boston, Massachusetts, United States